CLINICAL TRIAL: NCT00954746
Title: CORDLESS- Collagenase Optimal Reduction of Dupuytren's - Long-term Evaluation of Success Study
Brief Title: Longterm Observational Study in Subjects Treated With AA4500 in AUX-CC-854, 856, 857, 858 & 859
Status: Completed | Type: Observational
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: AUX-CC-860
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Dupuytren's Disease
Keywords: Advanced Dupuytren's Disease; Muscular Diseases; Musculoskeletal Diseases; Contracture Joint Diseases; Connective Tissue Diseases; Dupuytren's Contracture
MeSH Terms: conditions — Dupuytren Contracture; Muscular Diseases; Musculoskeletal Diseases; Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Follow-up: Subjects Previously Treated with AA4500

SUMMARY:
The purpose of study AUX-CC-860 is to assess the durability of response of the AA4500 treatment regimen. This study will also evaluate long-term safety and progression of disease in joints.

DETAILED DESCRIPTION:
Phase 3 non-treatment study in which Year 2 to Year 5 year follow-up of subjects who received AA4500 in the 9-month open-label studies (AUX-CC-854 and AUX-CC-856) or the 12-month double-blind with open-label extension studies (AUX-CC-857/AUX-CC-858 and AUX-CC-859). After completion of one of the above mentioned studies, subjects are enrolled and followed once a calendar year for 4 consecutive years with at least 6 months between consecutive visits.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study a subject had to:

* Have received at least one injection of AA4500 in one of the Auxilium sponsored studies (AUX-CC-854, AUX-CC-856, Studies AUX-CC-857/AUX-CC-858, or AUX-CC-859) and have at least one fixed-flexion contracture measurement after treatment with AA4500
* Be able and willing to comply with the yearly assessments outlined in the protocol, as determined by the investigator
* Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Advanced Dupuytren's Disease Previously Treated with AA4500 in Studies AUX-CC-854, AUX-CC-856, AUX-CC-857/AUX-CC-858, and AUX-CC-859
Sampling Method: Non-Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2009-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Contracture Measurements | yearly

SECONDARY OUTCOMES:
Immunogenicity, concomitant medications, medical history, and adverse events | yearly

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD, Study Director — Endo Health Solutions
Locations (39):
- United States (23):
  - Hope Research Institute, Phoenix, Arizona
  - Tucson Orthopedic Institute, P.C., Tucson, Arizona
  - Providence Clinical Research, Burbank, California
  - 100 UCLA Medical Plaza, Suite 305, Los Angeles, California
  - Hand Surgery Clinic, Palo Alto, California
  - The Hand and Upper Extremity Center of Georgia, P.C., Atlanta, Georgia
  - Southern Illinois Hand Center, S.C., Effingham, Illinois
  - Rockford Orthopedic Associates, Ltd., Rockford, Illinois
  - The Indiana Hand Center, Indianapolis, Indiana
  - Via Christi Research, Wichita, Kansas
  - Brigham and Women's Hospital, Department of Orthopedic Surgery, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Marquette General Health System, Marquette, Michigan
  - TRIA Orthopaedic Center, Minneapolis, Minnesota
  - Hospital for Special Surgery, New York, New York
  - SUNY Stony Brook - Department of Orthopedics, Stony Brook, New York
  - The Bone and Joint Center, Bismarck, North Dakota
  - Health Research Institute, Oklahoma City, Oklahoma
  - Hand Microsurgery & Reconstructive Orthopedics, Erie, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - University Orthopedics, Inc., Providence, Rhode Island
  - Alpha Clinical Research, Clarksville, Tennessee
  - Accurate Clincal Research, Houston, Texas
- Australia (6):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Rivercity Hospital, Auchenflower, Queensland
  - Caboolture Clinical Research Centre, Caboolture, Queensland
  - Peninsula Clinical Research, Kippa-Ring, Queensland
  - Menzies Research Institute, Hobart, Tasmania
  - Emeritus Research, Malvern, Victoria
- Denmark (3):
  - Gentofte Hospital, Hellerup, Copenhagen
  - Hospital of Aalborg, Aalborg
  - Rigshospitalet, Copenhagen
- Finland (2):
  - Dextra, Helsinki
  - Koskiklinikka, Tampere
- Sweden (2):
  - Department of Hand Surgery, Malmo
  - Department of Hand Surgery, Akademiska University Hospital, Uppsala
- United Kingdom (3):
  - Pulvertaft Hand Clinic, Derby, Derbyshire
  - Newcastle Biomedicine Clinical Research Facility, Newcastle, Newcastle Upon Tyne
  - Welsh Centre for Plastic Surgery Morriston Hospital, Swansea, Wales

REFERENCES:
- See also: Collagenase — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=009001121&QV1=COLLAGENASE
- See also: Dupuytren Society — http://www.dupuytren-online.info/